CLINICAL TRIAL: NCT04897581
Title: Establishing the Effectiveness of BBTI vs. PSR on Sleep and Pain Parameters in Adults With Musculoskeletal Orofacial Pain
Brief Title: BBTI vs PSR in Musculoskeletal Orofacial Pain Adults
Acronym: BBTI_PSR_21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ian Boggero, PhD (Other)
Responsible Party: Sponsor-Investigator, Ian Boggero, PhD, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65092
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Myofascial Pain; Myalgia
Keywords: local myalgia; centrally-mediated myalgia; masticatory pain; sleep; insomnia; behavioral therapy; self-regulation; depression; anxiety; fatigue
MeSH Terms: conditions — Myalgia; Sleep Initiation and Maintenance Disorders; Self-Control; Depression; Anxiety Disorders; Fatigue | interventions — phosphatidylserine receptor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data will be coded such that the Principal Investigator (PI) analyzing the data will be blind to conditions to prevent bias during the data collection and analysis. Also, the PI will remain blind through the study and will not provide either of the interventions. The statistician will be blind. The examiner will collect the data after de-identification of the sensitive and identifiable data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Therapy for Insomnia, BBTI (Experimental): Participants in this group will receive 3 sessions of BBTI over telehealth.
  Interventions: Behavioral: Brief Behavioral Therapy for Insomnia, BBTI
- Physical Self-Regulation, PSR (Experimental): Participants in this group will receive 3 sessions of PSR over telehealth.
  Interventions: Behavioral: Physical Self-Regulation, PSR

INTERVENTIONS:
Behavioral: Brief Behavioral Therapy for Insomnia, BBTI — BBTI includes sleep hygiene, stimulus control, and sleep restriction, and is administered in three 50-minute sessions over telehealth by psychologic team.
  Arms: Brief Behavioral Therapy for Insomnia, BBTI
Behavioral: Physical Self-Regulation, PSR — PSR is conducted over telehealth and consists of three 50-minute sessions focused on jaw relaxation exercises, proprioceptive awareness training, and diaphragmatic breathing entrainment.
  Arms: Physical Self-Regulation, PSR

SUMMARY:
This clinical study aims to compare the efficacy of two brief psychological interventions: Brief Behavioral Therapy for Insomnia (BBIT) and Physical Self-Regulation or (PSR) delivered over telehealth for the management of chronic musculoskeletal orofacial pain conditions (local myalgia, myofascial pain, centrally mediated myalgia) in a tertiary orofacial pain clinic. It is hypothesized that both interventions will produce beneficial changes and exploratory analysis will aim to establish which intervention -if any- is better for each specific outcome.

DETAILED DESCRIPTION:
New patients who come into the orofacial pain clinic are evaluated by a dental resident and given an orofacial pain diagnosis. If this primary diagnosis involves masticatory myofascial pain, local myalgia, or centrally-mediated myalgia, and if patients self-report poor sleep, they will be introduced to the study. An initial evaluation for PSR and BBTI will be scheduled over telehealth. If willing and eligible to participate, at the end of this first evaluation, they will be provided with an informed consent form and be randomly assigned to three sessions of PSR or three sessions of BBTI. After providing an e-consent, they will be sent a questionnaire battery on REDCap to assess their outcomes at pre-intervention. A REDCap daily questionnaire will be sent every day (morning and evening) starting one week before session 1 of the intervention, until two weeks after the last session. Moreover, to a small group of patients randomly selected, an actigraphy watch will be mailed. Two weeks after the last session of the intervention, a REDCap questionnaire will be sent to assess their outcomes at post-intervention. As per the current clinical protocol, all participants will be offered both interventions; only data from the first intervention will be utilized for the current study. All PSR and BBTI sessions will be conducted via telehealth using a HIPAA-compliant zoom account.

ELIGIBILITY:
Inclusion Criteria:

* present with a score on Insomnia Severity Index > 15
* have a primary diagnosis of chronic (onset more than 3 months before) MSK pain (myofascial pain and/or local myalgia and/or centrally mediated myalgia) from a board-certified orofacial pain specialist at UK Orofacial Pain Clinic
* maintain a stable medication regime in previous month and during the intervention
* older than 18 years old
* able to understand English
* willing to participate to telehealth intervention
* have internet access and an email address
* present with total STOP BANG score < 5

Exclusion Criteria:

* less than 18 years old
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Change in Self-report Insomnia Symptoms | At pre-intervention (1 week before starting with the intervention) and post-intervention (2 weeks after the last session of the intervention)
  Insomnia symptomatology will be assessed via the Insomnia Severity Index (ISI). The ISI includes seven items (sleep-onset, sleep maintenance, early morning awakening, satisfaction with current sleep pattern, interference with daily functioning, impairment attributed to sleep problems, distress caused by sleep problems), related to the prior 2 weeks on a five-point Likers scale (0= no problem, 4 = severe problem). The total score ranges from 0 to 28, with 28 indicating severe insomnia. The cut-off for the present study is 15. The ISI has good internal consistency and is demonstrated to be sensitive to changes in sleep of older adults following behavioral treatment for insomnia. Clinical improvement is defined as a reduction of ISI below the cut-off of 15.
Change in Self-report Average Pain Intensity | At pre-intervention (1 week before starting with the intervention), post-intervention (2 weeks after the last session of the intervention)
  The average pain intensity will be assessed using a Numeric Rating Scale (NRS) on a 10-point scale, where 0 coincides with "no pain" and 10 coincides with "worse pain ever felt".
Change in Self-report Quality of Life | At pre-intervention (1 week before starting with the intervention), post-intervention (2 weeks after the last session of the intervention)
  The overall quality of life will be assessed with 12-Item Short Form Health Survey (SF-12), a 12-item questionnaire designed to measure general health by addressing eight domains: limitations in social, physical, usual role activities because of physical health and emotional problems; bodily pain; general mental health; vitality; general health perceptions. SF-12 has been shown to reflect change over time like the long form SF-36 and to demonstrate good reliability and validity . Studies have addressed the impact of orofacial pain and sleep problems on health-related quality of life.
  The average score of the US population is set at 50. A score below this cut-off identifies a poor self-report quality of life.

SECONDARY OUTCOMES:
Change in Self-report Sleep Quality | At pre-intervention (1 week before starting with the intervention), post-intervention (2 weeks after the last session of the intervention)
  The sleep quality will be assessed via the RU-SATED, constituted by 6 items. RU-SATED appears to be a valid instrument for the assessment of sleep health among adults that is related to, but distinct from, other established sleep constructs. It provides a score from 0 to 12, with response to 6 questions. The lower the score, the worse the self-report sleep quality of the patient.
Sleep architecture | Each morning and each evening from the first session to 2 weeks after the last session of the intervention
  Sleep architecture will be assessed subjectively via daily morning and evening sleep diaries, sent to the participants via a REDCap survey. It will be assessed objectively via an actigraphy watch.
  The measured variables are sleep efficiency (SE), total sleep time (TST), sleep onset latency (SOL), number of awakening per night (NOA).
  For such variable, the change in outcomes will be collected; therefore, there is not a scale for measuring the change.
Change in Self-report Depression Symptoms | At pre-intervention (one week before the first session of the intervention), at post-intervention (two weeks after the last session of the intervention) and every day during the intervention period
  Depression symptoms will be assessed at pre- and post-intervention via Pain-Health Questionnaire-4 (PHQ4). The Pain-Health Questionnaire (PHQ, 4 items) allows for a brief and accurate measurement of signs/symptoms of anxiety and depression, by providing an overall measure of symptom burden, as well as functional impairment and disability with a 4-point scale . PHQ-4 has demonstrated strong psychometric properties and have been validated for use in the general population. The first two questions of PHQ4 (PHQ-2) consists of core criteria for depression. The score goes from 0 to 4 for each question (for a total of 8, being 8 the most severe depression symptoms), and a score of 3 or above on the Depression subscale represent a reasonable cut off point for identifying potential cases of depression and a psychologist or counselor referral will be offered.
  Depression symptoms will be also monitored daily via morning and evening daily diaries, sent to the participant via a REDCap survey. �
Change in Self-report Anxiety Symptoms | At pre-intervention (one week before the first session of the intervention), at post-intervention (two weeks after the last session of the intervention) and every day during the intervention period
  Anxiety symptoms will be assessed at pre- and post-intervention via Pain-Health Questionnaire-4 (PHQ4). The Pain-Health Questionnaire (PHQ, 4 items) allows for a brief and accurate measurement of signs/symptoms of anxiety and depression, by providing an overall measure of symptom burden, as well as functional impairment and disability with a 4-point scale. PHQ-4 has demonstrated strong psychometric properties and have been validated for use in the general population. The last two questions (GAD-2) consists of core criteria for anxiety, with score going from 0 (no symptoms) to 4 (most severe anxiety symptoms) for each question. A score of 3 or above on the Anxiety subscale represents a reasonable cut off point for identifying potential cases of depression and a psychologist or counselor referral will be offered.
  Anxiety and depression symptoms will be also monitored daily via morning and evening daily diaries, sent to the participant via a REDCap survey. �
Change in Self-report Headache Intensity | At pre-intervention (one week before the first session of the intervention), at post-intervention (two weeks after the last session of the intervention)
  Headache measures will investigate the severity of headache on a 10-point scale (Numeric Rating Scale, NRS), with 0 identifying "no pain", and 10 identifying "the worst pain experienced".
Change in Self-report Headache Frequency | At pre-intervention (one week before the first session of the intervention), at post-intervention (two weeks after the last session of the intervention)
  This questionnaire investigate headache disability (in terms of lack of productivity, missing working days or school days), frequency and intensity will be also assessed using the Migraine Disability Assessment Test (MIDAS, 6-item).
  Each item identifies the total number of days per month of headache frequency (being 0 "no days of headache" and being 30 "each day with headache"). The minimum score is 0, the maximum is 150, with the upper limit identifying the highest frequency of headaches.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Boggero, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
The data will be de-identified from the sensible data information. The data will be retained for 5 years after the end of the study. There is no intension to share the IPD with other researchers.
  However, the data collected from this study will be utilised by the investigators for possible future studies.

REFERENCES:
- [Background] Ballou S, Katon J, Rangan V, Cheng V, Nee J, Iturrino J, Lembo A. Brief Behavioral Therapy for Insomnia in Patients with Irritable Bowel Syndrome: A Pilot Study. Dig Dis Sci. 2020 Nov;65(11):3260-3270. doi: 10.1007/s10620-020-06182-w. Epub 2020 Mar 9. PMID 32152868